CLINICAL TRIAL: NCT05037851
Title: A Randomized Controlled Open-label Study to Assess the Safety and Tolerability of Nebulized PC945 for Prophylaxis or Pre-emptive Therapy Against Pulmonary Aspergillosis in Lung Transplant Recipients (OPERA-S Study)
Brief Title: A Safety Study of PC945 (Opelconazole) Prophylaxis or Pre-emptive Therapy Against Pulmonary Aspergillosis in Lung Transplant Recipients (OPERA-S Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PC_ASP_007
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Aspergillosis
MeSH Terms: conditions — Pulmonary Aspergillosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, active-controlled, parallel-group multi-center study
Masking Description: The study will be an open-label study. For the purposes of the exploratory efficacy assessments, however, the Data Review Committee determining the presence of pulmonary fungal disease will be blinded as to treatment assignment. The Sponsor will limit knowledge of treatment assignment to as few sponsor personnel as possible to reduce bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Opelconazole (Experimental): 14.8 mg opelconazole administered twice daily for 12 weeks
  Interventions: Drug: Opelconazole
- Standard of Care (SoC) (Active Comparator): Mold-active SoC prophylaxis/pre-emptive therapy
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Opelconazole — Nebulizer suspension
  Other Names: PC945
  Arms: Opelconazole
Drug: Standard of Care — Standard of Care
  Arms: Standard of Care (SoC)

SUMMARY:
A study to evaluate the safety and tolerability of opelconazole for the prevention of fungal aspergillus infections in the lung in participants who have received a lung transplant.

DETAILED DESCRIPTION:
Part 1 of the study comprises a 12 week Prophylaxis or Pre-emptive Therapy Phase. Part 2 comprises a 4-week Safety Follow-Up Phase.

The study will screen single or double lung transplant recipients due to receive a mold-active antifungal: either as de novo prophylaxis or as pre-emptive therapy (for participants with Aspergillus spp. colonization of the respiratory tract but no evidence of pulmonary fungal disease). Only participants who fulfill all the inclusion and none of the exclusion criteria will be randomized.

ELIGIBILITY:
Key Inclusion Criteria:

2. Participant has received either a single or double lung transplant but did not receive any other organ transplant (e.g., heart, kidney, etc.) at the time of the lung transplantation. History of prior transplant (>1 year) is acceptable

6a. (De novo prophylaxis immediately post transplant): participant must be ready to be randomized and start anti-mold prophylaxis within 72 hours of returning to the intensive care unit (ICU) after the transplant surgery or

6b. (Pre-emptive therapy): participant must meet all of the following:

* Aspergillus spp. colonization of the respiratory tract confirmed within 91 days (13 weeks) after a lung transplant. Colonization is defined according to the 2010 International Society for Heart Lung Transplantation (ISHLT) Consensus Statement definition criteria for colonization
* Without evidence of pulmonary fungal disease
* Must be ready to start anti-mold medication within 96 hours after the positive culture(s), galactomannan or polymerase chain reaction (PCR) result(s) were reported

Key Exclusion Criteria:

1. Participant would normally receive nebulized amphotericin B as the only mold active antifungal agent as initial SoC prophylaxis or pre-emptive therapy
2. Fungal disease requiring systemic antifungal treatment at the time of transplant
3. Has received a mold active antifungal agent post-transplant (Note: a participant who receives a mold active antifungal agent within 24 hours before, during, or after the transplant procedure will not be excluded if the mold active medication was stopped within 72 hours of returning to the ICU after the transplant surgery, or prior to randomization (whichever happens first)
4. Has previously received opelconazole
5. Is receiving, or who is due to receive at any time during the study, an investigational medicinal agent
6. Is participating, or who is due to participate at any time during the study, in a therapeutic clinical trial. For any other trials (e.g. observational or using approved medication), consultation with Pulmocide and the medical monitor is required.
7. Has an endobronchial stent in situ
8. Known history of allergy, hypersensitivity, or any previous serious reaction to any component of the opelconazole formulation, azoles, echinocandins, or amphotericin B
9. Elevated alanine transaminase (ALT) or, aspartate transaminase (AST) > 5 x the upper limit of normal (ULN)
10. Any known history or current evidence of alcohol or drug abuse that, in the Investigator's opinion, would exclude the participant from participation in the study

12. Life expectancy is not expected to be sustained for the duration of the trial (16 weeks), in the opinion of the investigator

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete 12 weeks of therapy | Baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Clinical Development, Study Director — Pulmocide Ltd
Locations (18):
- United States (16):
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, La Jolla, California
  - Clinical Research Site, Los Angeles, California
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Tampa, Florida
  - Clinical Research Site, Maywood, Illinois
  - Research Site, St Louis, Missouri
  - Clinical Research Site, New York, New York
  - Clinical Research Site, The Bronx, New York
  - Clinical Research Site, Philadelphia, Pennsylvania
  - Clinical Research Site, Pittsburgh, Pennsylvania
  - Clinical Research Site, Nashville, Tennessee
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site 1, Houston, Texas
  - Clinical Research Site 2, Houston, Texas
  - Clinical Research Site 3, Houston, Texas
- Canada (2):
  - Clinical Research Site, Edmonton
  - Clinical Research Site, Toronto

IPD SHARING:
Plan to Share IPD: No